CLINICAL TRIAL: NCT05973149
Title: Tolerance, Safety, Pharmacokinetics, and Preliminary Anti-tumor Activity of QLH12016 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Trial of QLH12016 in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLH12016-101
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLH12016 dose escalation (Experimental): Daily dosages are predetermined by Safety Monitoring Committee after the initial starting dose cohort at the end of Cycle 1 (each cycle is 28 days)
  Interventions: Drug: QLH12016
- QLH12016 in mCRPC with specific biomarkers (Experimental): Daily dosage and schedule at a recommended Phase 2 dose based on data from Arm A
  Interventions: Drug: QLH12016
- QLH12016 in mCRPC without specific biomarkers (Experimental): Daily dosage and schedule at a recommended Phase 2 dose based on data from Arm A
  Interventions: Drug: QLH12016
- QLH12016 in less pretreated mCRPC (Experimental): Daily dosage and schedule at a recommended Phase 2 dose based on data from Arm A
  Interventions: Drug: QLH12016

INTERVENTIONS:
Drug: QLH12016 — according to the scheme description

SUMMARY:
To evaluate the tolerance, safety, pharmacokinetics, and preliminary anti-tumor activity of QLH12016 in patients with metastatic castration resistant prostate cancer

DETAILED DESCRIPTION:
Subjects will use QLH12016 for the treatment of mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign a written informed consent form
2. Male, aged ≥ 18 years
3. ECOG：0-1
4. Expected survival time of at least 3 months
5. Prostate adenocarcinoma confirmed by histological or cytological without neuroendocrine or small cell characters
6. Continuous treatment with luteinizing hormone releasing hormone analogue or luteinizing hormone releasing hormone antagonist (drug castration), or previous bilateral orchiectomy (surgical castration); Subjects who did not receive bilateral orchiectomy must plan to maintain effective luteinizing hormone releasing hormone analog or luteinizing hormone releasing hormone antagonist treatment throughout the study period
7. testosterone≤50 ng/dL or 1.7 nmol/L
8. CRPC is defined as the occurrence of one or more of the following three events in a subject while undergoing castration treatment: ① PSA progression, defined as at least two increases in PSA levels (PSA value>1 ng/mL, interval of at least 1 week, consecutive 2 times, increase>50% from baseline); ② Disease progression as defined in RECIST v1.1; ③ The progression of skeletal diseases as defined by the PCWG3 standard, where bone scans reveal ≥ 2 or more new lesions
9. Metastatic lesion with imaging evidence. At least one target lesion exists
10. Received 1-2 lines of new endocrine therapy (such as enzalutamide, abiolone, etc.) after developing castration resistance（ArmA-C）
11. Received 0-1 line chemotherapy treatment (such as docetaxel) during the hormone sensitive period and the castration resistance period（ArmA-C）
12. Arm B: with specific biomarkers; Arm C: without specific biomarkers; Arm D: received 0 or 1 line of new endocrine therapy, and no chemotherapy during hormone sensitive and castration resistant stages
13. The functional level of important organs must meet the following requirements (no blood components, hematopoietic stimulating factors, cell growth factors, leukemic drugs, platelet enhancing drugs, etc. are allowed to be used within 7 days before obtaining laboratory examination): Absolute neutrophil count ≥ 1.5 × 10^9/L; Platelets ≥ 100 × 10^9/L; Hemoglobin ≥ 100 g/L; Serum albumin ≥ 30 g/L; AST and ALT ≤ 2.5 × Upper limit of normal reference value (ULN), if accompanied by liver metastasis, ALT and AST ≤ 5 × ULN; Total bilirubin ≤ 1.5 × ULN (Gilbert syndrome≤ 3 × ULN); Serum creatinine ≤ 1.5 × ULN, if >1.5 × ULN, then the creatinine clearance rate (CLcr) ≥ 50 mL/min; LVEF>50%
14. Effective contraceptive measures from signing the informed consent to 90 days after the last use of the study drug
15. Recover from all AEs of previous anti-cancer treatment (i.e. ≤ grade 1, according to CTCAE v5.0), excluding alopecia (any grade) and peripheral sensory nerve ≤ grade 2, hypomagnesemia or lymphocytopenia, as well as other abnormalities that the benefit of receiving treatment is greater than the risk

Exclusion Criteria:

1. Metastasis of the central nervous system (CNS), leptomeningeal metastasis or spinal cord compression caused by metastasis (exceeding the physiological alternative dose) requiring hormone treatment
2. Radiation therapy that has irradiated more than 25% of the bone marrow was performed within 4 weeks. Palliative radiation therapy is allowed to alleviate pain caused by bone metastasis during the study period
3. Treatment with similar drugs
4. Received other clinical trial drugs or major surgeries within 4 weeks (sufficient wound healing after major surgeries must undergo clinical evaluation)
5. Systemic anti-cancer treatment within the first 2 weeks (bicalutamide, Mitomycin C or Nitroso urea 6 weeks, enzalutamide 5 weeks, and abiolone 4 weeks). Medications that maintain castration are allowed.
6. Planned bilateral orchiectomy during the study treatment
7. Inability to swallow, chronic diarrhea and bowel obstruction, or other factors affecting drug administration and absorption
8. Epilepsy or disease that can induce seizure within 12 months (including a history of transient ischemic attack, stroke, brain trauma with disorders of consciousness, etc.)
9. History of psychotropic substance abuse, alcoholism, or drug use, neurological or mental disorders, including dementia or hepatic encephalopathy
10. Any of the following conditions occurs within 12 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure (New York Heart Association III or IV), cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism or other thromboembolic diseases with clinical significance
11. Any of the following conditions within 6 months: congenital long QT syndrome, torsade de pointes ventricular tachycardia, arrhythmia (including persistent ventricular tachyarrhythmia and Ventricular fibrillation), left anterior half block (double vessel block) or persistent arrhythmia above NCI-CTCAE grade 2, Atrial fibrillation of any level (in the case of Asymptomatic isolated Atrial fibrillation, grade ≥ 2)
12. Cardiovascular diseases under poor control, including angina pectoris, pulmonary hypertension or serious cardiac rhythm or conduction abnormalities
13. QTcF>450 ms
14. Active, uncontrolled bacterial, fungal, or viral infections, including but not limited to: 1) Active hepatitis B virus (HBV), hepatitis C virus (HCV) infected persons (hepatitis B surface antigen [HBsAg] positive or hepatitis B core antibody [HBcAb] positive, HBV DNA virus copy number ≥ 500 IU/mL, HCV antibody positive and HCV RNA higher than the detection limit of the analysis method); 2) Syphilis required treatment; 3) History of congenital immunodeficiency or organ transplantation, or HIV (HIV) positive
15. Clinically uncontrollable third space effusion, such as pleural effusion, peritoneal effusion, pericardial effusion, etc. that cannot be controlled by drainage or other measures and cannot be included in the group according to the judgment of the investigator
16. Other malignant tumors within 5 years (excluding cured basal cell skin cancer, papillary thyroid cancer, etc.)
17. Concomitant diseases seriously endangering the safety of the subject or affect the completion of the study, such as hypertension (systolic pressure ≥ 160 mmHg and/or diastolic pressure ≥ 100 mmHg) that cannot be controlled by two or more antihypertensive drugs, diabetes not well controlled, etc
18. History of hypertensive crisis or hypertensive encephalopathy
19. Allergy to any study drug component
20. Gastrointestinal perforation, gastrointestinal or non gastrointestinal fistula, or abdominal abscess within 6 months
21. Any life-threatening bleeding event within 3 months, including the need for blood transfusion treatment, surgery or local treatment, and continuous medication treatment
22. Subjects who may increase research related risks, interfere with the interpretation of research results, or are deemed unsuitable for inclusion by the researcher

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Arm A： Incidence of Dose Limiting Toxicities | 28 Days
  First Cycle Dose limiting toxicities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug
Arm A：Maximum Tolerated Dose | 28 Days
  The Maximum Tolerated Dose determined by the Incidence of Dose Limiting Toxicities
Arm A：Recommended Phase 2 Dose | 28 Days
  Recommended Phase 2 Dose determined by the frequency of Incidence of Dose Limiting Toxicities
Arm A：AE | 20 weeks
  The incidence, severity and correlation with the study drug of adverse events (AEs) evaluated according to the National Cancer Institute (NCI) - General Terminology of Adverse Events (CTCAE) Version 5.0
Arm A：SAE | 20 weeks
  The incidence, severity and correlation with the study drug of Serious adverse event (SAE) evaluated according to the National Cancer Institute (NCI) - General Terminology of Adverse Events (CTCAE) Version 5.0
Arm B-D：PSA Response Rate | 20 weeks
  a decrease of ≥ 50% in PSA levels from baseline to baseline, and reassessed PSA relief after ≥ 3 weeks in each arm
Arm B-D：Objective Response Rate | 20 weeks
  the percentage of "CR/PR" subjects in each arm

SECONDARY OUTCOMES:
Cmax | 20 weeks
  The highest plasma drug concentration
Tmax | 20 weeks
  The time blood drug concentration reaching Cmax
AUC | 20 weeks
  The area enclosed by the drug time curve and the time axis
Arm A：ORR | 20 weeks
  the percentage of "CR/PR" subjects
Arm A：PSA Response Rate | 20 weeks
  a decrease of ≥ 50% in PSA levels from baseline to baseline, and reassessed PSA relief after ≥ 3 weeks
Arm B-D：AE | 20 weeks
  The incidence, severity and correlation with the study drug of adverse events (AEs) evaluated according to the National Cancer Institute (NCI) - General Terminology of Adverse Events (CTCAE) Version 5.0
Arm B-D：SAE | 20 weeks
  The incidence, severity and correlation with the study drug of Serious adverse event (SAE) evaluated according to the National Cancer Institute (NCI) - General Terminology of Adverse Events (CTCAE) Version 5.0
DOR | 20 weeks
  The time between the initial evaluation of CR or PR and disease progression
DCR | 20 weeks
  the percentage of "CR/PR/SD" subjects
rPFS | 20 weeks
  The time between the first administration of the investigational drug and the first recording of disease progression (determined according to RECIST v1.1 and PCWG3) or the date of all-cause death (whichever occurs first)
OS | 20 weeks
  The time between the first trial drug administration and patient death due to various reasons

OTHER OUTCOMES:
Biomarkers | 20 weeks
  Using next-generation sequencing，reverse transcription DNA and quantitative polymerase chain reaction to evaluate tumor mutational burden and other signal pathway indicators

CONTACTS AND LOCATIONS:
Overall Officials: Zhisong He, Phd, Principal Investigator — Department of Urology, Peking University First Hospital; Hongqian Guo, Phd, Principal Investigator — Department of Urology, Drum Tower Hospital, Nanjing University School of Medicine
Locations (2):
- China (2):
  - Department of Urology, Peking University First Hospital, Beijing, Beijign
  - Department of Urology, Drum Tower Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No